CLINICAL TRIAL: NCT04146805
Title: A Phase 1a, Double Blind, Placebo-Controlled, Single-Center, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability Pharmacokinetics, and Pharmacodynamics of BLD-0409 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BLD-0409 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-0409-101
Record Dates: First submitted 2019-10-23; First posted 2019-10-31 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-02

CONDITIONS: Chronic Liver Disease; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1SAD/Part 2 MAD:Active Treatment(BLD-0409) (Experimental): For each cohort in both study parts, 6 subjects will be randomized to active (BLD-0409). Study drug will be administered orally once a day, with an option to evaluate twice daily dosing (BID) in Part 2 MAD cohort(s)
  Interventions: Drug: BLD-0409
- Part 1SAD/Part 2 MAD:Control(Matched Placebo) (Placebo Comparator): For each cohort in both study parts, 2 subjects will be randomized to control (matched placebo). Study drug will be administered orally once a day, with an option to evaluate twice daily dosing (BID) in Part 2 MAD cohort(s).
  Interventions: Drug: Control: Placebo

INTERVENTIONS:
Drug: BLD-0409 — For each cohort in both study parts, 8 subjects will be randomized in a 6:2 ratio to active (BLD-0409) : control (matched placebo). Study drug will be administered orally once a day, with an option to evaluate twice daily dosing (BID) in Part 2 MAD cohort(s).
  Arms: Part 1SAD/Part 2 MAD:Active Treatment(BLD-0409)
Drug: Control: Placebo — Subjects will be randomized in a 6:2 ratio to control (matched placebo). Study drug will be administered orally once a with an option to evaluate twice daily dosing (BID) in Part 2 MAD cohort(s).
  Arms: Part 1SAD/Part 2 MAD:Control(Matched Placebo)

SUMMARY:
A Phase 1a, Double Blind, Placebo-Controlled, Single-Center, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability Pharmacokinetics, and Pharmacodynamics of BLD-0409 in Healthy Volunteers

DETAILED DESCRIPTION:
The study will evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses (SAD) and multiple ascending doses (MAD) of BLD-0409 in healthy volunteers (HV) to facilitate the dose/dosing regimen selection for future clinical studies with BLD-0409 in various chronic liver diseases.

The study consists of two parts:

Part 1: SAD in HV with up to 6 cohorts (including a food effect cohort). For SAD cohorts and planned dosing schedule.

Part 2: MAD over 14 days with up to 6 cohorts. For MAD cohorts and planned dosing schedule.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be included in the study only if all the following criteria apply:

Age and Gender

1. Male and female subjects 18-55 years of age (inclusive) at the time of signing the PICF.

   Diagnosis and disease characteristics
2. Subjects must be in good general health, in the opinion of the Investigator, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of study drug.
3. Subjects must have clinical laboratory values within normal ranges or < 1.2 times upper limit of normal (ULN) as specified by the testing laboratory, unless deemed not clinically significant (NCS) by the Investigator, with exception of liver function tests which cannot be above the ULN.
4. Body mass index (BMI) 18 to ≤ 32 kg/m2. Reproductive Considerations Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. For details refer to Appendix 4.
5. Female subjects and female partners of male subjects must use double barrier contraception and refrain from oocyte donation from first dose of study drug and for 60 days after last dose of study drug. Estrogen-containing products are not allowed.
6. Male subjects must agree to use highly effective, double barrier contraception and refrain from sperm donation from first dose of study drug and for 90 days after last dose of study drug.
7. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. Females not of childbearing potential must be surgically infertile or post-menopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by follicle-stimulating hormone (FSH) level > 40 mIU/mL at Screening.

   Informed Consent
8. Subjects must provide signed informed consent prior to study entry and have the ability and willingness to attend and comply with the necessary visits at the study site.

Exclusion Criteria

Subjects meeting ANY of the following exclusion criteria are NOT eligible to be randomized into the study:

Medical Conditions

1. Recent (less than 6 weeks) wound, or presence of an ongoing non-healing skin wound.
2. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will complete the study per protocol.
3. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia.
4. Serious local or systemic infection within 1 month of Screening requiring antibiotic treatment or history of recurrent infections.
5. Surgery within the past 3 months prior to the first study drug administration determined by the Investigator to be clinically relevant.

   Diagnostic Assessments
6. Positive for human immunodeficiency virus (HIV) antibody or antigen.
7. Positive hepatitis C virus (HCV) antibody or positive hepatitis B surface antigen (HBsAg).
8. Systolic blood pressure (BP) > 150 mmHg or < 90 mmHg or diastolic BP > 90 mmHg or < 50 mmHg at Screening with one repeat allowed per the Investigator's discretion at Screening and Day -1.
9. Heart rate < 40 beats per minute (bpm) or > 100 bpm at Screening.
10. Prolonged QTcF (>450 ms for males and >470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting ECG, as judged by the Investigator.
11. Females with heavy menstruating cycles and borderline-low iron studies. Prior Therapy
12. All prescription and over the counter medications (including herbal medications), except for non-estrogen contraceptives, are prohibited within 7 days prior to the first study drug administration and throughout the entire duration of the study.
13. Any estrogen-containing products, e.g., contraceptives, patch, cream, implants within 14 days prior to the first study drug administration.

    Prior/Concurrent Clinical Study Experience
14. Administration of investigational product in another study within 30 days prior to the first study drug administration, or five half-lives, whichever is longer.

    Other Exclusions
15. Significant weight loss or gain between Screening and first study drug administration.
16. Blood donation or significant blood loss within 60 days prior to the first study drug administration.
17. Plasma donation within 7 days prior to the first study drug administration.
18. Females who are pregnant or breastfeeding.
19. Diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior first study drug administration.
20. History or presence of alcohol or drug abuse (including recreational marijuana use) within the 1 year prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period.
21. Positive urine drug screen/alcohol breath test at Day -1 (admission). Repeat urine drug screens will be permitted for suspected false positive results.
22. Intake of alcohol or caffeine-containing products from 48 hours before first study drug administration.
23. Active smokers and users of nicotine-containing products.
24. Failure to satisfy the Investigator of fitness to participate for any other reason.

Lifestyle Considerations Meals and Dietary Restrictions

1. Subjects will fast from all food and drink except water for ≥ 10 hours before morning study drug administration on Day 1.
2. Except during the periods of fasting, standard meals and snacks will be provided at the discretion of the Investigator while subjects are confined in the study site.
3. For food effect Cohort 1e:

   1. On Day 8, subjects will be provided a standard high calorie breakfast from 30 minutes before dose administration (and to be consumed entirely within that 30 minutes). The meal is to follow United States Food and Drug Administration (FDA) guidance regarding caloric content and composition. The test meal should derive approximately 150, 250 and 500 600 calories from protein, carbohydrate, and fat, respectively. An example test meal would be two eggs fried in butter, two strips of bacon, and two slices of toast with butter, four ounces of hash brown potatoes and eight ounces of whole milk. Substitutions in this test meal can be made as long as the meal provided a similar amount of calories from protein, carbohydrate and fat and has comparable meal volume and viscosity. Vegetarians may be enrolled provided that there is a consultation with a dietician regarding comparable calories, volume and viscosity.
   2. Water restrictions may be needed. No water is allowed 1 hour before and after dosing, after which time, water is allowed ad libitum.
4. Subjects will refrain from consumption of Seville oranges, grapefruit or grapefruit juice, from 48 hours before the start of study drug until after the final PK sample is obtained.
5. Subjects will refrain from diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior to dosing on Day 1.

Caffeine, Alcohol, and Tobacco

1. During each dosing session, subjects will abstain from ingesting caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) for 48 hours before the start of dosing until after collection of the final pharmacokinetic (PK) and/or pharmacodynamic sample.
2. During each dosing session, subjects will abstain from alcohol for 48 hours before the start of dosing until EOS visit.
3. Active smokers and users of nicotine-containing products will be excluded from the study.

Other Restrictions Subjects will avoid strenuous physical activity (e.g. weightlifting, running, bicycling) from 24 hours prior to Day 1 until discharge from the study site and for 24 hours prior to the EOS visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | up to 56 days
  AEs will be assessed by determining the incidence, severity, and dose relationship of adverse events
Number of subjects with treatment-related subjects changes in physical examinations | up to 56 days
  Assessed by performing physical examinations include general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes, from baseline by dose, through out the study.
  Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of treatment subjects with treatment-related changes in heart rate | up to 56 days
  Assessed by collecting and evaluating any observed changes in heart rate. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of treatment subjects with treatment-related changes in systolic & diastolic blood pressure | up to 56 days
  Assessed by collecting and evaluating any observed changes in systolic & diastolic blod pressure. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of treatment subjects with treatment-related changes in body temperature | up to 56 days
  Assessed by collecting body temperature using a thermometer. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in ECG tracings | up to 56 days
  Assessed by performing 12-lead ECGs, and evaluating ECG tracings from baseline, by dose. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in QTc intervals | up to 56 days
  Assessed by performing 12-lead ECGs, and evaluating QTc intervals from baseline, by dose. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in hematology clinical laboratory test results. | up to 56 days
  Assessed by collecting and analyzing subjects' blood from baseline by dose. Results in subjects dosed with BLD-0409 treatment will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in chemistry clinical laboratory test results. | up to 56 days
  Assessed by collecting and analyzing subjects' blood from baseline by dose. Results in subjects dosed with BLD-0409 treatment will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in urinalysis clinical laboratory test results. | up to 56 days
  Assessed by collecting and analyzing subjects' urine from baseline by dose. Results in subjects dosed with BLD-0409 treatment will be compared to those dosed with placebo.
Number of subjects with treatment-related changes in serology clinical laboratory test results. | up to 56 days
  Assessed by collecting and analyzing subjects' blood from baseline by dose. Results in subjects dosed with BLD-0409 treatment will be compared to those dosed with placebo.

SECONDARY OUTCOMES:
Area under the drug concentration-time curve from time zero to the last measurable concentration (AUClast) | up to 56 days
  To characterize the Plasma pharmacokinetics(PK) of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo
Area under the drug concentration time curve from time 0 to infinity (AUC0-inf) | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Maximum observed drug concentration (Cmax) | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Time of the maximum drug concentration (tmax) | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Apparent terminal elimination rate constant (kel) | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Apparent elimination half life (t½) | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Apparent oral clearance | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Apparent terminal volume of distribution | up to 56 days
  To characterize the Plasma PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Amount excreted during each collection interval (Ae(t'-t'')) | up to 56 days
  To characterize the urine PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Total amount of drug excreted unchanged in the urine over the entire period of sample collection | up to 56 days
  To characterize the urine PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Percentage of dose excreted unchanged during each collection interval (Fe(t' t")) and over the entire period of sample collection | up to 56 days
  To characterize the urine PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Renal clearance (CLr) for each collection interval and over the entire period of sample collection | up to 56 days
  To characterize the urine PK of BLD-0409 in healthy volunteers. Results in subjects dosed with BLD-0409 will be compared to those dosed with placebo.
Any observed Changes in serum Lysophosphatidic Acid Receptor (LPA) C18:2 | up to 56 days
  Measured by serum in subjects dosed with BLD-0409 will be compared to those dosed with placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No